CLINICAL TRIAL: NCT04349917
Title: Large-scale Brain Organization During Cognitive Control in ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-0112; R00MH102349 (NIH)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: methylphenidate; functional connectivity; graph theory; cognitive control
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Sugars

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover design. Each subject with ADHD participates in two sessions, one on drug and one on placebo (order randomized ). Both subjects and experimenters are blind to the order.
Who Masked: Participant, Investigator
Masking Description: The pharmacy that provides the drug/placebo works from a randomized subject order defining whether each subject received drug first or placebo first. Only the pharmacists know this order, and the drug and placebo look identical to the participants and the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo, then Methylphenidate (Placebo Comparator): All children with ADHD in this study will receive one dose of methylphenidate and one dose of placebo over the course of two sessions approximately one week apart (order randomized and double-blind).
  Interventions: Drug: Methylphenidate; Other: Placebo
- Methylphenidate, then Placebo (Experimental): All children with ADHD in this study will receive one dose of methylphenidate and one dose of placebo over the course of two sessions approximately one week apart (order randomized and double-blind).
  Interventions: Drug: Methylphenidate; Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — A single, low dose of methylphenidate (0.3 mg/kg) will be administered on the drug day.
  Other Names: Ritalin
Other: Placebo — A matching placebo pill will be administered on the placebo day.
  Other Names: Sugar pill

SUMMARY:
The purpose of this study is to test whether children with attention-deficit/hyperactivity disorder (ADHD) are impaired in the ability to flexibly adapt brain network organization in response to shifting cognitive demands during the exertion of cognitive control, by assessing changes in network dynamics resulting from stimulant administration in children with ADHD, and how those changes relate to behavioral and symptom improvements. Subjects will be children with ADHD aged 8-12. Subjects will participate in multiple testing sessions that include: diagnosis and eligibility screening, neuropsychological and behavioral testing, and, if eligible, MRI scans and a medication challenge. Children with ADHD who are enrolled in the medication challenge will undergo one MRI scan on placebo and one MRI scan on stimulant medication, counterbalanced and double-blind. Functional connectivity will be measured using functional MRI and innovative graph theoretical analytic tools will be implemented. Network metrics will be related to symptomatology and behavioral testing measures. It is hypothesized that stimulant administration in children with ADHD will increase flexibility in network reconfiguration in response to changing cognitive control demands as compared to when they are on placebo. It is further hypothesized that the degree to which brain network organization is changed will be related to the degree of improvement in cognitive control performance.

ELIGIBILITY:
Inclusion Criteria:

* Between 8-12 years old
* Diagnosis of ADHD (for ADHD group); ADHD group only can have comorbid Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnoses of oppositional defiant disorder, conduct disorder, depressive disorders, or anxiety disorders
* ADHD subjects must never have been treated with medication for their ADHD

Exclusion Criteria:

* Wechsler Intelligence Scale for Children-Fifth Edition Full-Scale Intelligence Quotient (IQ) < 80
* Wechsler Individual Achievement Test-Third Edition Word Reading < 85
* Any neurologic or developmental disabilities
* Any reading or learning disabilities
* Visual impairment that cannot be corrected-to-normal
* Color blindness
* Documented hearing impairment greater than 25 decibels (dB) loss in either year
* Have already gone through puberty (Tanner Stage II or higher)
* Medical contraindication to MRI
* Any psychoactive medication

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Cohen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between December 2016 and March 2020.
Pre-assignment Details: A total of 47 participants were screened during a behavioral visit. Of those not randomized, 8 did not meet inclusion criteria and 2 withdrew from study.
Groups:
- Methylphenidate, Then Placebo: Participants received a single, low dose of methylphenidate (0.3 mg/kg) before the first MRI scan. Approximately one week later, participants received a matching placebo pill before the second MRI scan.
- Placebo, Then Methylphenidate: Participants received a matching placebo pill before the first MRI scan. Approximately one week later, participants received a single, low dose of methylphenidate (0.3 mg/kg) before the second MRI scan.
Period: First Intervention (2-4 Hours)
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methylphenidate
Started | 19 | 18
Received Intervention | 19 | 17
Completed | 19 | 16
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unable to Swallow Pill | 0 | 1
Period: Washout Period (4-20 Days)
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methylphenidate
Started | 19 | 16
Completed | 19 | 16
Not Completed | 0 | 0
Period: Second Intervention (2-4 Hours)
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methylphenidate
Started | 19 | 16
Received Intervention | 19 | 16
Completed | 19 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate, Then Placebo | Placebo, Then Methylphenidate | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.71 (0.92) | 9.75 (1.41) | 9.73 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 14 | 31
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Resting State Brain Network Organization
Description: Assessment of network topology during a resting state using functional connectivity estimates. Modularity will be determined by applying graph theoretical methods to functional connectivity estimates acquired during functional magnetic resonance imaging (fMRI) scans. Modularity is measured on a -1 to 1 scale, with higher scores indicating stronger community structure, or a stronger tendency of clusters of brain regions to separate into distinct, highly interconnected networks with sparse connections across networks. The optimal modularity value depends on the context. For example, during complex tasks lower modularity is better, while during basic, automatic tasks higher modularity is better.
Time Frame: 1 to 3 hours after administration of intervention
Population: Participants excluded due to excessive head motion (mean framewise displacement (FD) > 0.5mm or fewer than 150 timepoints remaining after scrubbing all timepoints with FD > 0.2mm), incomplete brain coverage, or poor-quality fMRI data. Participants must have good data from both methylphenidate and placebo scan days to be included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methylphenidate: Participants received a single, low dose of methylphenidate (0.3 mg/kg) before MRI scan
- Placebo: Participants received a matching placebo pill before MRI scan.
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale | 0.223 (0.026) | 0.228 (0.034)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Test type: Superiority; p = 0.532, t-test, 2 sided

2. Primary Outcome: Task-Based Brain Network Organization
Description: Assessment of network topology during the Go/No-go (GNG) regular and GNG reward tasks. Subjects see a series of sports balls and are told to respond to most balls (go trials), but not to some specific balls (no-go trials). GNG tasks are identical, except in the rewarded task, correct fast go responses and correct withholding on no-go trials are rewarded with 1 cent and 5 cents respectively. Graph theoretical methods are applied to functional connectivity estimates from fMRI scans to determine modularity during each task. Modularity (-1 to 1 scale) measures the degree to which the whole-brain system separates into distinct communities, such that greater modularity reflects stronger community structure, or stronger tendency of brain regions to separate into distinct, highly interconnected networks with few connections across networks. Optimal modularity value depends on context. During complex tasks lower modularity is better, while higher modularity is better for basic tasks.
Time Frame: 1 to 3 hours after administration of intervention
Population: Participants excluded due to excessive head motion (mean framewise displacement [FD] > 0.5mm or fewer than 150 timepoints remaining after scrubbing all timepoints with FD > 0.2mm), incomplete brain coverage, or poor-quality fMRI data. Participants must have good data from both methylphenidate and placebo scan days to be included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale
  GNG regular | 0.213 (0.041) | 0.218 (0.040)
  GNG reward | 0.235 (0.051) | 0.213 (0.055)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Analysis for GNG regular task; Test type: Superiority; p = 0.579, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Analysis for GNG reward task; Test type: Superiority; p = 0.034, t-test, 2 sided

3. Primary Outcome: Rest-Task Reconfiguration
Description: Assessment of reconfiguration of network topology between the GNG regular task and the resting state and GNG reward task and resting state. In the GNG tasks, subjects see a series of sports balls and are told to respond to most of the balls (go trials), but not to some specific balls (no-go trials). GNG tasks are identical, except in the rewarded task, correct fast go responses and correct withholding on no-go trials are rewarded with 1 cent and 5 cents respectively. Normalized mutual information will be determined by applying the same graph theoretical methods to functional connectivity estimates acquired during fMRI scans for each rest-task pair. Normalized mutual information is measured on a 0 to 1 scale, with higher scores indicating more similarity in network structure across task and rest conditions.
Time Frame: 1 to 3 hours after administration of intervention
Population: Participants excluded due to excessive head motion (mean framewise displacement [FD] > 0.5mm or fewer than 150 timepoints remaining after scrubbing all timepoints with FD > 0.2mm), incomplete brain coverage, or poor-quality fMRI data. Participants must have good data from both scan days and all tasks being compared to be included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  GNG regular | 0.104 (0.055) | 0.119 (0.058)
  GNG reward | 0.122 (0.074) | 0.150 (0.074)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Analysis for reconfiguration between rest and GNG regular task; Test type: Superiority; p = 0.296, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Analysis for reconfiguration between rest and GNG reward task; Test type: Superiority; p = 0.169, t-test, 2 sided

4. Primary Outcome: Drug-induced Normalization
Description: Assessment of how changes in brain network topology relate to improvements in behavioral performance on the GNG regular and reward tasks, in which subjects respond to go stimuli and withhold responses to no-go stimuli. GNG tasks are identical, except subjects are rewarded for good performance on the reward task. Brain measures include change in modularity during rest, GNG regular, and GNG reward (Outcome Measures 1, 2); behavioral measures include change in commission rate, omission rate, and coefficient of variation of response time during GNG tasks (Outcome Measures 5-7). Pearson correlations are used to relate change in brain measures with change in behavioral measures from the placebo to the methylphenidate scans. Positive correlations indicate that subjects with greater change in the brain measure had greater change in the behavioral measure. Negative correlations indicate that subjects with less change in the brain measure had greater change in the behavioral measure.
Time Frame: 1 to 3 hours after administration of intervention
Population: Participants excluded due to excessive head motion (mean framewise displacement [FD] > 0.5 mm or fewer than 150 timepoints remaining after scrubbing all timepoints with FD > 0.2 mm), incomplete brain coverage, or poor-quality fMRI data. Participants excluded if incomplete behavioral GNG data. Must have good data from both scan days to be included.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Methylphenidate and Placebo: Participants received a single, low dose of methylphenidate (0.3 mg/kg) before one MRI scan and a matching placebo pill before a separate MRI scan.
Arm/Group | Methylphenidate and Placebo
Number analyzed (Participants) | 18
correlation coefficient
  Delta rest mod vs delta GNG reg commission rate | -0.361 [-0.693 to 0.097]
  Delta rest mod vs delta GNG reg omission rate | 0.508 [0.084 to 0.776]
  Delta rest mod vs delta GNG reg RT variability | 0.287 [-0.178 to 0.647]
  Delta rest mod vs delta GNG rew commission rate | 0.162 [-0.303 to 0.564]
  Delta rest mod vs delta GNG rew omission rate | -0.224 [-0.606 to 0.243]
  Delta rest mod vs delta GNG rew RT variability | 0.003 [-0.440 to 0.445]
  Delta GNG reg mod vs delta GNG reg commission rate | -0.033 [-0.468 to 0.416]
  Delta GNG reg mod vs delta GNG reg omission rate | -0.170 [-0.570 to 0.271]
  Delta GNG reg mod vs delta GNG reg RT variability | -0.195 [-0.587 to 0.271]
  Delta GNG rew mod vs delta GNG rew commission rate | 0.220 [-0.246 to 0.604]
  Delta GNG rew mod vs delta GNG rew omission rate | -0.276 [-0.640 to 0.189]
  Delta GNG rew mod vs delta GNG rew RT variability | -0.027 [-0.464 to 0.420]
Statistical Analysis 1: Comparison: Methylphenidate and Placebo; Change in rest modularity vs change in GNG regular commission rate; Test type: Superiority; p = 0.118, Pearson correlation
Statistical Analysis 2: Comparison: Methylphenidate and Placebo; Change in rest modularity vs change in GNG regular omission rate; Test type: Superiority; p = 0.022, Pearson correlation
Statistical Analysis 3: Comparison: Methylphenidate and Placebo; Change in rest modularity vs Change in GNG regular RT Variability; Test type: Superiority; p = 0.220, Pearson correlation
Statistical Analysis 4: Comparison: Methylphenidate and Placebo; Change in rest modularity vs change in GNG reward commission rate; Test type: Superiority; p = 0.496, Pearson correlation
Statistical Analysis 5: Comparison: Methylphenidate and Placebo; Change in rest modularity vs change in GNG reward omission rate; Test type: Superiority; p = 0.343, Pearson correlation
Statistical Analysis 6: Comparison: Methylphenidate and Placebo; Change in rest modularity vs change in GNG reward RT variability; Test type: Superiority; p = 0.988, Pearson correlation
Statistical Analysis 7: Comparison: Methylphenidate and Placebo; Change in GNG regular modularity vs change in GNG regular commission rate; Test type: Superiority; p = 0.892, Pearson correlation
Statistical Analysis 8: Comparison: Methylphenidate and Placebo; Change in GNG regular modularity vs change in GNG regular omission rate; Test type: Superiority; p = 0.473, Pearson correlation
Statistical Analysis 9: Comparison: Methylphenidate and Placebo; Change in GNG regular modularity vs Change in GNG regular RT Variability; Test type: Superiority; p = 0.409, Pearson correlation
Statistical Analysis 10: Comparison: Methylphenidate and Placebo; Change in GNG reward modularity vs change in GNG reward commission rate; Test type: Superiority; p = 0.351, Pearson correlation
Statistical Analysis 11: Comparison: Methylphenidate and Placebo; Change in GNG reward modularity vs change in GNG reward omission rate; Test type: Superiority; p = 0.238, Pearson correlation
Statistical Analysis 12: Comparison: Methylphenidate and Placebo; Change in GNG reward modularity vs Change in GNG reward RT Variability; Test type: Superiority; p = 0.909, Pearson correlation

5. Secondary Outcome: Go/No-go (GNG) Commission Rate
Description: Evaluation of commission errors assessed during the GNG regular and GNG reward tasks. In the GNG tasks, subjects see a series of sports balls and are told to respond to most of the balls (go trials), but not to some specific balls (no-go trials). GNG tasks are identical, except in the rewarded task, correct fast go responses and correct withholding on no-go trials are rewarded with 1 cent and 5 cents respectively. In both tasks, commission errors occur on trials on which participants respond to a stimulus ("go" response) when they are supposed to withhold a response ("no-go" trial). Commission errors are scored from 0 (no commission errors) to 1 (100% commission errors), with lower values indicating better performance.
Time Frame: 1 to 3 hours after administration of intervention
Population: Participants must have good data from both methylphenidate and placebo scan days to be included in this analysis. Participants included if they completed at least one task.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale
  GNG regular | 0.396 (0.213) | 0.403 (0.206)
  GNG reward | 0.292 (0.176) | 0.348 (0.181)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Analysis for GNG regular task; Test type: Superiority; p = 0.806, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Analysis for GNG reward task; Test type: Superiority; p = 0.003, t-test, 2 sided

6. Secondary Outcome: Go/No-go (GNG) Omission Rate
Description: Evaluation of omission errors assessed during the GNG regular and GNG reward tasks. In the GNG tasks, subjects see a series of sports balls and are told to respond to most of the balls (go trials), but not to some specific balls (no-go trials). GNG tasks are identical, except in the rewarded task, correct fast go responses and correct withholding on no-go trials are rewarded with 1 cent and 5 cents respectively. In both tasks, omission errors occur on trials on which participants do not respond to a "go" stimulus to which they are supposed to respond. Omission errors are scored from 0 (no omission errors) to 1 (100% omission errors), with lower values indicating better performance.
Time Frame: 1 to 3 hours after administration of intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale
  GNG regular | 0.071 (0.116) | 0.104 (0.119)
  GNG reward | 0.040 (0.055) | 0.101 (0.111)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Analysis for GNG regular task; Test type: Superiority; p = 0.093, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Analysis for GNG reward task; Test type: Superiority; p = 0.0001, t-test, 2 sided

7. Secondary Outcome: Go/No-go (GNG) Response Time Variability
Description: Evaluation of response time variability assessed during the GNG regular and GNG reward tasks. In the GNG tasks, subjects see a series of sports balls and are told to respond to most of the balls (go trials), but not to some specific balls (no-go trials). GNG tasks are identical, except in the rewarded task, correct fast go responses and correct withholding on no-go trials are rewarded with 1 cent and 5 cents respectively. Coefficient of variation (standard deviation / mean) will be calculated for response time in GNG regular and GNG reward tasks separately to account for group differences in mean response time.
Time Frame: 1 to 3 hours after administration of intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 33 | 33
coefficient of variation
  GNG regular | 0.298 (0.104) | 0.344 (0.155)
  GNG reward | 0.253 (0.071) | 0.342 (0.146)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Analysis for GNG regular task; Test type: Superiority; p = 0.075, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Analysis for GNG reward task; Test type: Superiority; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the First Intervention through 24-48 hours following the Second Intervention, an overall total of between 5-22 days depending on the length of the Washout Period (Washout Period range: 4-20 days).
Description: Safety Population includes all participants who received at least one dose of intervention
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 11/35 | 9/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=35) | Placebo (N=36)
Heart Racing (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Stomachache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 7 | 4
Increased Energy (General disorders) | 0 | 1
Change in Appetite (Metabolism and nutrition disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Changes in Mood (Psychiatric disorders) | 4 | 1
Difficulty Falling Asleep (Psychiatric disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04349917/Prot_SAP_000.pdf